CLINICAL TRIAL: NCT06731491
Title: Terapias Complementares no Processo de Envelhecimento de Pessoas Vivendo Com HIV: Uma Abordagem Multi-design Sobre o Efeito da Massoterapia, Aromaterapia e do exercício físico
Brief Title: Complementary Therapies in the Aging Process of People Living With HIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital das Clínicas, University of Sao Paulo Medical School (Unknown); Ministry of Education, Brazil (Other Government)
Responsible Party: Principal Investigator, Andre Pereira dos Santos, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAAE:78708524.5.0000.5659
Record Dates: First submitted 2024-11-18; First posted 2024-12-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: HIV; aging; concurrent training; people living with hiv; massage
MeSH Terms: interventions — Exercise; Massage; Aromatherapy

STUDY DESIGN:
Intervention Model Description: Non-Randomized and Blinded Parallel Cross-Sectional Clinical Study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Control Group (No Intervention): There will be no intervention and group participants will be advised to maintain their routine as normal.
- G1 (Experimental): Intervention Group - Concurrent Training for People Living with HIV who have been on Antiretroviral Therapy for 10 years or more
  Interventions: Other: Concurrent Training
- G2 (Experimental): Intervention Group - Concurrent Training for People Living with HIV who have been on Antiretroviral Therapy for less than 10 years
  Interventions: Other: Concurrent Training
- G3 (Experimental): Intervention Group - Concurrent Training for People Living with HIV who have been on Antiretroviral Therapy for less than 10 years and had CD4/CD8 < 1
  Interventions: Other: Concurrent Training
- G4 (Experimental): Intervention Group - Massage Therapy for People Living with HIV who have been on Antiretroviral Therapy for 10 years or more
  Interventions: Other: Massage therapy and Aromatherapy
- G5 (Experimental): Intervention Group - Massage Therapy for People Living with HIV who have been on Antiretroviral Therapy for less than 10 years
  Interventions: Other: Massage therapy and Aromatherapy
- G6 (Experimental): Intervention Group - Massage Therapy for People Living with HIV who have been on Antiretroviral Therapy for less than 10 years and have CD4/CD8 < 1
  Interventions: Other: Massage therapy and Aromatherapy

INTERVENTIONS:
Other: Concurrent Training — Strength and aerobic training in the same training session for a period of 12 weeks, 3 times a week and with an average training time of 60 minutes
  Other Names: exercise; training
  Arms: G1; G2; G3
Other: Massage therapy and Aromatherapy — Massage Therapy with Aromatherapy twice a week for a period of 12 weeks and an average time of 40 minutes per session.
  Other Names: massage
  Arms: G4; G5; G6

SUMMARY:
PROBLEM DELIMITATION AND JUSTIFICATION Complementary therapies, including physical exercise and massage therapy, are ways to mitigate the side effects of aging, HIV infection and ART. In parallel, there are studies that seek to propose a way to analyze muscle strength and endurance, balance, walking ability, body composition, immunological, metabolic and biochemical parameters, sarcopenia, frailty syndrome, sleep quality, self-perception of health, self-esteem, perception of body image, anxiety, depression, cognitive function, medication adherence, quality of life, diet and level of physical activity in people living with HIV (PLWH). However, the impact of concurrent training, massage therapy and aromatherapy on these parameters together in PLWH with different times of diagnosis and consequences of the low CD4/CD8 ratio during their clinical history has not yet been investigated.

RELEVANCE Understanding the impact of concurrent training, massage therapy and aromatherapy, as complementary therapies, on physical, biochemical and psychosocial parameters according to the time of diagnosis and consequences of the low CD4/CD8 ratio is a way to evaluate the effect of these interventions on different profiles of the same population, and consequently, favor the development of other studies that can propose training and massage for PLWH, considering the time of diagnosis and the impact of HIV on their body.

GENERAL OBJECTIVE To evaluate the impact of complementary therapies on variables associated with the aging of people living with HIV, considering the time of diagnosis and the CD4/CD8 ratio.

Study design The research project has a multidesign characteristic, that is, different study designs will be used that communicate with each other to provide a broad approach to the effect of complementary therapies on the aging process of PLWH. The study designs used will be: systematic review and meta-analysis, cross-sectional observational study, and blinded clinical trial.

Intervention protocol The kinetics of heart rate and oxygen consumption, peak running speed (Vpeak), running speed at the ventilatory threshold, and respiratory exchange ratio will be assessed before and after the 12-week intervention. In addition, the estimated maximum load (1RM) in strength training will be verified in exercises for the upper limbs: front pulldown, bench press on the machine, and lateral elevation of the shoulders with dumbbells; and lower limbs: leg press 90°, adductor and abductor chair, and plantar flexion on the bench before and after the 12-week intervention. Massage and aromatherapy sessions will be performed once a week for 12 weeks for 30 minutes in the dorsal region. The massage protocol that will be used includes classic massage movements (superficial sliding, deep sliding, friction, rolling, kneading) with grape seed vegetable oil mixed with lavender essential oils, being a 2% mixture (50 drops of essential oil for 100ml of vegetable oil).

Statistical analysis In this project, the variables considered as independent are concurrent training and relaxing massage with the use of essential oils. An initial exploratory analysis will be performed to check the distribution behavior of the data. If the data present a normal distribution, a descriptive analysis (measures of central tendency, SD, CI) of the outcome variables in the periods (pre- and post-intervention) will be performed. If there is no normal distribution of the data, the description of the outcome variables will occur through median, minimum and maximum value, and 25th and 75th interquartile range.

If there is a normal distribution of the data, the t-test for dependent samples will be used to identify differences in the pre- and post-intervention period for the intervention and control groups. Subsequently, the one-way ANOVA will be used to verify differences between the intervention and control groups, in the pre- and post-intervention period. If there is no normal distribution, the Mann-Whitney U test for dependent samples will be used to identify differences in the pre- and post-intervention period for the intervention and control groups. Subsequently, the Wilcoxon test for independent samples will be used to verify differences between the intervention and control groups, in the pre- and post-intervention period. It is not the objective of this project to compare the effect of the intervention between concurrent training and relaxing massage with the use of essential oils. The effect size (η2) of concurrent training and relaxing massage with the use of essential oils on the outcome variables will be calculated. The analyses will be performed in SPSS 23.0 software, assuming prior statistical significance (α = 0.05).

DETAILED DESCRIPTION:
PROBLEM DELIMITATION AND JUSTIFICATION Complementary therapies, including physical exercise and massage therapy, are ways to mitigate the side effects of aging, HIV infection and ART. In parallel, there are studies that seek to propose a way to analyze muscle strength and endurance, balance, walking ability, body composition, immunological, metabolic and biochemical parameters, sarcopenia, frailty syndrome, sleep quality, self-perception of health, self-esteem, perception of body image, anxiety, depression, cognitive function, medication adherence, quality of life, diet and level of physical activity in people living with HIV (PLWH). However, the impact of concurrent training, massage therapy and aromatherapy on these parameters together in PLWH with different times of diagnosis and consequences of the low CD4/CD8 ratio during their clinical history has not yet been investigated.

RELEVANCE Understanding the impact of concurrent training, massage therapy and aromatherapy, as complementary therapies, on physical, biochemical and psychosocial parameters according to the time of diagnosis and consequences of the low CD4/CD8 ratio is a way to evaluate the effect of these interventions on different profiles of the same population, and consequently, favor the development of other studies that can propose training and massage for PLWH, considering the time of diagnosis and the impact of HIV on their body.

GENERAL OBJECTIVE To evaluate the impact of complementary therapies on variables associated with the aging of people living with HIV, considering the time of diagnosis and the CD4/CD8 ratio.

Specific objectives

In adults living with HIV:

1. Conduct a systematic review of the literature with the purpose of compiling scientific evidence addressing the effects of concurrent training on a variety of variables, including sleep quality, self-perception of health, self-esteem, quality of life, perception of body image, anxiety, depression, cognitive function, medication adherence, anthropometric measurements, immunological and metabolic parameters, biomarkers associated with aging, body composition, motor function and frailty.
2. Conduct a systematic review of the literature to compile scientific evidence related to the effects of massage therapy with the use of essential oils on the following variables: sleep quality, self-perception of health, self-esteem, quality of life, perception of body image, anxiety, depression, cognitive function, medication adherence, as well as immunological and metabolic parameters.
3. Investigate the occurrence of frailty syndrome in adults living with HIV, considering temporal variables related to HIV diagnosis and the implications of the low CD4/CD8 ratio.
4. To evaluate the impact of concurrent training through pre- and post-intervention determination and comparative analyses on a wide range of variables, including sleep quality, self-perception of health, self-esteem, quality of life, perception of body image, anxiety, depression, cognitive function, medication adherence, anthropometric measurements, immunological and metabolic parameters, biomarkers associated with aging, body composition, motor function and frailty. This examination will be carried out according to the times of HIV diagnosis and the consequences associated with the low CD4/CD8 ratio.
5. To evaluate the effect of massage therapy with the use of essential oils in adults living with HIV, analyzing variables such as sleep quality, self-perception of health, self-esteem, quality of life, perception of body image, anxiety, depression, cognitive function, medication adherence, as well as immunological and metabolic parameters. This evaluation will be carried out considering the times of HIV diagnosis and the implications of the low CD4/CD8 ratio.

Study design The research project has a multidesign characteristic, that is, different study designs will be used that communicate with each other to provide a broad approach to the effect of complementary therapies on the aging process of PLWH. The study designs used will be: systematic review and meta-analysis, cross-sectional observational study, and blinded clinical trial.

Intervention protocol The kinetics of heart rate and oxygen consumption, peak running speed (Vpeak), running speed at the ventilatory threshold, and respiratory exchange ratio will be assessed before and after the 12-week intervention. In addition, the estimated maximum load (1RM) in strength training will be verified in exercises for the upper limbs: front pulldown, bench press on the machine, and lateral elevation of the shoulders with dumbbells; and lower limbs: leg press 90°, adductor and abductor chair, and plantar flexion on the bench before and after the 12-week intervention. Massage and aromatherapy sessions will be performed once a week for 12 weeks for 30 minutes in the dorsal region. The massage protocol that will be used includes classic massage movements (superficial sliding, deep sliding, friction, rolling, kneading) with grape seed vegetable oil mixed with lavender essential oils, being a 2% mixture (50 drops of essential oil for 100ml of vegetable oil).

Concurrent training The concurrent training will consist of a warm-up phase (a 5-minute light-to-moderate walk), followed by 40 minutes of strength training using free weights and machines to work the body's main muscle groups, and 20 minutes of aerobic training, controlling heart rate reserve (HR) on a treadmill. Finally, there will be a 5-minute cool-down phase (active stretching). The training program will be performed 3 times a week for 12 weeks, totaling 36 training sessions. The periodization was based on the guidelines of the American College of Sports Medicine.

For strength training, the movement cadence will be 1 second and 2 seconds for the concentric and eccentric phases, respectively. The time interval between each exercise will be between 90-120 seconds.

The intervention will be performed at LaCiDH of EEFERP/USP. The aerobic training load will be adjusted using HRres, calculated using the following equation:

HRres = [(HRmax - HRrest) x intensity] + HRrest

The resting heart rate will be assessed before the prescription of aerobic exercise and at the end of the fourth and eighth weeks for load adjustment. Participants will remain at rest in a chair for 10 minutes to record their HR, and then their HR will be taken to calculate their resting HR. The maximum heart rate (HRmax) will be calculated using the equation proposed by Tanaka et al.

The initial load for strength training will be determined during the first week of the intervention protocol. The load will be adjusted until it corresponds to 10-12 maximum repetitions for each exercise. Load adjustments will occur weekly and will be performed as follows: during the last weekly training session, participants will be instructed to perform 10 (first 8 weeks) or 8 repetitions (9th week onwards) in the first set for each exercise, and as many repetitions as possible before concentric failure in the last set of each exercise. For each repetition greater than 10 (first 8 weeks) or 8 (9th week onwards), 1 kg will be added for lower limb exercises and 0.5 kg for upper limb exercises. This increase will be incorporated into the following training session the following week.

Monitoring of concurrent training Before each training session, measurements of blood pressure, HR and blood oxygen saturation (SpO2) will be taken, following the standards of the SBC, SBH and SBN (57) and SBPT (58). The measurements will be taken using a stethoscope and aneroid sphygmomanometer of the "Premium®" brand, a heart rate monitor of the "Polar FT7®" brand and a digital oximeter of the "Oximeter®" brand. In the absence of contraindicated vital signs, the training protocol will be carried out. Additionally, the HR and BP of the participants will be monitored throughout the training period.

Relaxing massage using essential oils 12 sessions of relaxing massage and aromatherapy will be carried out, lasting 30 minutes, on the back of the trunk. The intensity of the pressure of the relaxing massage will be moderate, which corresponds to the pressure exerted on the vulva of the sphygmomanometer between 50 and 80 mmHg. The massage will be performed by two professionals with experience in performing the massage and applying the pressure necessary to stimulate the relaxing massage. A mixture of grape seed oil and lavender essential oil will be used.

Data collection Data will be collected by collecting information from the research participant, including anamnesis and questionnaires that assess sleep quality, self-perception of health, self-esteem, quality of life, perception of body image, anxiety, depression, cognitive function and adherence to medication therapy. In addition, some anthropometric measurements will be taken. This information will be collected by the research team. Routine laboratory tests - to assess immunological and metabolic parameters, and biochemical variables associated with aging - will be performed by laboratory technicians from HC-FMRP/USP. The analysis of multicompartmental body composition by Dual Energy X-ray Absorptiometry (DXA) to estimate fat mass, lean mass, and bone mineral density will be performed by prior appointment by a radiology technician responsible for operating the equipment at LaCiDH of EEFERP/USP. Motor tests to estimate maximum load in concurrent training exercises, handgrip strength, isokinetic knee extension muscle strength, and gait will be evaluated at LaCiDH of EEFERP/USP. Balance will be evaluated at the Laboratory of Biomechanics and Motor Control of EEFERP/USP. Aerobic variables will be verified at the Laboratory of Exercise Physiology and Metabolism (LAFEM) of EEFERP/USP.

Statistical analysis In this project, the variables considered as independent are concurrent training and relaxing massage with the use of essential oils. An initial exploratory analysis will be performed to check the distribution behavior of the data. If the data present a normal distribution, a descriptive analysis (measures of central tendency, SD, CI) of the outcome variables in the periods (pre- and post-intervention) will be performed. If there is no normal distribution of the data, the description of the outcome variables will occur through median, minimum and maximum value, and 25th and 75th interquartile range.

If there is a normal distribution of the data, the t-test for dependent samples will be used to identify differences in the pre- and post-intervention period for the intervention and control groups. Subsequently, the one-way ANOVA will be used to verify differences between the intervention and control groups, in the pre- and post-intervention period. If there is no normal distribution, the Mann-Whitney U test for dependent samples will be used to identify differences in the pre- and post-intervention period for the intervention and control groups. Subsequently, the Wilcoxon test for independent samples will be used to verify differences between the intervention and control groups, in the pre- and post-intervention period. It is not the objective of this project to compare the effect of the intervention between concurrent training and relaxing massage with the use of essential oils. The effect size (η2) of concurrent training and relaxing massage with the use of essential oils on the outcome variables will be calculated. The analyses will be performed in SPSS 23.0 software, assuming prior statistical significance (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age ≥ 50 years
* Diagnosed with HIV at age ≥ 18 years
* HIV diagnosis for > 6 months
* Use of ART with unchanged medication for > 6 months
* Clinically stable, with undetectable viral load (< 40 copies per ml of blood)
* Not undergoing treatment for opportunistic diseases or cancer
* Maintaining stable body weight (less than 10% variation in the past six months)
* No musculoskeletal disorders impairing the ability to perform exercise (e.g., - --- Duchenne Muscular Dystrophy and Becker Muscular Dystrophy)
* Medical clearance for physical exercise
* Not using medications that could significantly alter body composition (e.g., testosterone, growth hormone, and insulin-like growth factor 1)
* Not pregnant
* Not breastfeeding
* Not using prosthetics
* No amputations of any body part
* Not engaged in a regular physical exercise program in the past six months

Exclusion Criteria:

* Showing any symptoms that would contraindicate their continued participation in the training program, or that would result in risks due to the practice of exercises
* Showing concurrent diseases, classified as (1) infections (Mycobacterium Avium, Cytomegalovirus, Pneumocystis Carinii Pneumonia, Herpes Simplex Virus, Tuberculosis, Toxoplasmosis); (2) neoplasms (Kaposi's Sarcoma, Non-Hodgkin's Lymphoma, Hodgkin's Lymphoma), (3) autoimmune diseases (Autoimmune Hemolytic Anemia)
* Declining participation in the study
* Failing to complete all stages of the study, including the minimum of 80% attendance at training sessions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  Quantifying masses: visceral and subcutaneous fat, lean and bone, detecting values for the total body and by segments (upper limbs, trunk, lower limbs and head) using kg and % of total weight as units of measurement.
Biomarkers associated with aging | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The biomarkers will be: IL-1β, IL-2, IL-10, IL-12, IL-17A, IL-18, IFN-γ, cIAP, XIAP, Caspase 3, Caspase 8, Caspase 9, TGFβ-1, BAX protein, TNF-α, IL-6, hsCRP and PBMC: prelamin-A, p16INK4a, p21WAF-1, p53 and activated phospho-p53, sCD14 (unit/ml)
Quality of sleep | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  Sleep quality will be assessed before and after interventions using the validated Pittsburgh Sleep Quality Index (PSQI) questionnaire for Brazil. The PSQI measures sleep quality retrospectively over the previous month using self-report/recall. It consists of nineteen individual items that assess seven components of sleep quality: (1) sleep duration; (2) sleep disturbance; (3) sleep latency; (4) daytime dysfunction due to sleepiness; (5) sleep efficiency; (6) overall sleep quality; and (7) use of sleep medications. These seven-component scores (scored from 0 to 3) are summed to produce a global score between 0 and 21, with higher scores indicating poorer sleep quality. A global PSQI score ≤5 indicates good sleep quality and >5 indicates poor sleep quality. PSQI has demonstrated good psychometric performance in Brazil.
Handgrip Strength Measurement | From the start of recruitment to the end of the interventions there will be approximately 15 weeks.
  Three attempts will be made on the dominant hand, with one-minute intervals between them, and the highest measurement in kg will be recorded.
Mobility Performance | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The test is performed by walking at the highest speed for 6 minutes. The result will be obtained from the number of meters walked during the test.
Frailty syndrome assessment | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  Questions will be asked to assess the five components of the Frailty Phenotype, proposed by Fried. Participants with three or more impairments in these components will be classified as frail, and those with one or two, as pre-frail. Those with all negative tests for the components of the frailty phenotype will be considered robust or non-frail.
Knee extension muscle strength in isokinetic | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The knee extension test will be performed with five repetitions, considering the peak torque value of the concentric contraction in the unit newton per meter (Nm) for recording
Gait assessment | The time between the start of recruitment and the end of the interventions will be approximately 15 weeks.
  The gait assessment will be performed using the Timed Up and Go (TUG) test. The evaluator starts the timing when the participant stands up, and stops only when the participant is sitting in the chair with their arms and torso supported. The time recorded is recorded in seconds.
Balance assessment | The period from the start of recruitment to the end of the interventions will be approximately 15 weeks.
  The Berg Balance Scale will be used to assess balance. It consists of 14 items related to balance and postural control. The total score is 56 points and, depending on the score, it is possible to determine whether balance is impaired (0-20), acceptable (21-40) or good (41-56).
Self-perception of health | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  To assess self-perceived health, two questions from the WHOQOL-HIV-Bref will be used. This is an abbreviated instrument developed by the World Health Organization (2003) to assess the quality of life of people living with HIV and validated in Brazil. It consists of 31 questions to assess six domains (Physical, Psychological, Level of Independence, Social Relationships, Environment and Spirituality) and the overall state of quality of life and health perception. Five responses are possible on a Likert scale with values from one to five. The score ranges from 4 to 20, with higher scores indicating better quality of life.
Self-esteem | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  Self-esteem will be assessed using the Rosenberg self-esteem scale, validated in Brazil. The scale has 10 sentences, 6 referring to positive self-image and self-worth, and the other 4 referring to negative self-image or self-deprecation. Three Likert-style scores are possible: "I agree," "I neither agree nor disagree," and "I disagree," and the higher the score on the scale, the higher the level of self-esteem.
Quality of Life and Health Perception | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The WHOQOL-HIV-Bref, an instrument developed by the World Health Organization (2003) to assess the quality of life of people living with HIV, has been validated in Brazil. It consists of 31 questions to assess six domains (Physical, Psychological, Level of Independence, Social Relationships, Environment and Spirituality) and the overall state of quality of life and health perception. Five responses are possible on a Likert scale with values from one to five, the score ranges from 4 to 20, and higher scores indicate better quality of life.
Perception of body image | From the start of recruitment to the end of the interventions will be approximately 15 weeks.
  Body image perception will be assessed using the Stunkard silhouette assessment scale, adapted and validated for Brazil, in which a series of silhouettes with a given value are presented to participants so that they can indicate the one that most resembles their current body perception and the silhouette they consider ideal. Subsequently, the size and shape currently perceived are compared with the size and shape considered ideal, using the value of the indicated silhouettes, subtracting the value considered ideal from the current value. The result ranges from -8 to 8 and indicates the discrepancy score that reveals the level of dissatisfaction with body image, with zero being the value for satisfaction with body image and values other than zero being dissatisfaction with body image.
Anxiety and Depression | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The Hospital Anxiety and Depression Scale (HAD) by Zigmond and Snaith, which has been validated in Brazil. The scale consists of 14 questions, seven of which assess anxiety (HADS-A) and seven assess depression (HADS-D). The score for each subscale ranges from 0 to 21 points, and the cutoff score for determining anxiety or depression is greater than or equal to nine points.
Cognitive function | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  MOCA- Montreal Cognitive Assessment - Cognitive screening questionnaire that investigates the following factors: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall and orientation. It is also validated in Brazil. The questionnaire consists of specific sections for each factor, totaling 30 points. In addition, it is possible to add one point if the assessed person's years of schooling are ≤ 12 years.
Medication adherence | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The "Cuestionario para la Evaluación de la Adhesión al Tratamiento Antiretroviral" (CEAT-VIH), by Remo, validated in Brazil, will be used to assess adherence to drug therapy. It is a self-administered instrument with 20 questions. The score is given by the sum of all items and ranges from a minimum of 17 to 89 points; the higher the score, the greater the drug adherence.

SECONDARY OUTCOMES:
Immunological parameters | From the beginning of recruitment until the end of the interventions will be approximately 15 weeks.
  To verify the clinical stability of the volunteers, the amount of viral load (copies/mL) and the count of TCD4+ lymphocytes (cells/mm³) and TCD8 (cells/mm³) will be checked. The viral load level will be considered detectable when HIV RNA is > 40 copies mL-1. Viral load will be determined by the Abbott Real Time method, using the Siemens - Versant® HIV-1 RNA 3.0 kit and DNA Analyzer System 340® device. The TCD4+ and TCD8 lymphocyte count (cells/mm³) will be performed by Flow Cytometry, using the Multitest® kit and the Facs Calibur® cytometer.
Body weight | From the beginning of recruitment until the end of the interventions will be approximately 15 weeks.
  The measurements will be performed using an electronic anthropometric scale by Filizola®, (Personal model for up to 180 kg, Campo Grande, MS). The participant will stand on the scale platform wearing as little clothing as possible (shorts - males, and shorts and top - females), with their arms extended along the body in a static position. Body weight will be recorded in kilograms (kg) with an accuracy of 100 grams (g). The body weight measured on the scale will only be used to insert data used in the DXA adjustment.
Determination of Maximum Strength (1RM) | From the beginning of recruitment to the end of the interventions there will be approximately 15 weeks.
  The participants' maximum strength, considered as the ability to lift a certain weight in a single repetition (1RM), will be assessed at two times: pre- and post-intervention, following the maximum repetition test (RM) procedures described in the literature by Brzycki (1993). The RM will be: 1RM = Weight lifted (kg)/[1.0278-(0.0278 x number of repetitions)]
Physical activity level | From the start of recruitment to the end of the interventions will be approximately 15 weeks.
  The Brazilian version of the International Physical Activity Questionnaire - Short Version (IPAQ-SV) will be applied to measure the level of physical activity. The IPAQ-SV groups and conceptualizes the categories as follows: (a) Sedentary: does not perform any physical activity for at least 10 continuous minutes during the week; (b) insufficiently active: practices physical activities for at least 10 continuous minutes per week, but not enough to be classified as active. (c) Active - meets the following recommendations: (a) vigorous physical activity: ≥ 3 days/week and ≥ 20 min/session; (b) moderate activity or walking: ≥ 5 days/week and ≥ 30 min/session; (c) any added activity: ≥ 5 days/week and ≥ 150 min/week. (d) Very active - meets the following recommendations: (a) vigorous activity: ≥ 5 days/week and ≥ 30 min/session; (b) vigorous activity: ≥ 3 days/week and ≥ 20 min/session + moderate activity and/or walking ≥ 5 days/week and ≥ 30 min/session.
Energy intake | From the beginning of recruitment to the end of the interventions there will be approximately 15 weeks.
  Three 24-hour food recalls will be performed over a period of one week (2 weekdays and 1 weekend day), where detailed information about meals will be recorded, generally from the day before the participant's assessment. The food intake data obtained in household measurements (coffee spoon, tea spoon, ladle, cups, plates, etc.) will be converted to an estimate in grams and milliliters in order to enable the chemical analysis of food consumption processed by the Dietpro® nutritional analysis program, version 5i. The software will allow the insertion of foods reported by the participant, not yet available in the program, assigning nutritional values according to the Brazilian Food Composition Table (TACO) and USDA - National Nutrient Database for Standard Reference. The average energy and macronutrient consumption (as a % of the total caloric value) of the three days will be considered for the dietary assessment.
Peak Oxygen Consumption (VO2peak) | From the start of recruitment to the end of the interventions will be approximately 15 weeks.
  Participants will perform an incremental test to exhaustion on a treadmill (T170; Cosmed, Rome, Italy) to analyze VO2peak and peak running speed (Vpeak). The test will begin at a speed at which the participant feels comfortable walking for 10 minutes (the speed will be adjusted if necessary during this period). After establishing the ideal speed for 10 minutes, the speed will remain stable until the end of the test and the treadmill incline will be increased by 1% every 3 minutes until voluntary exhaustion. VO2 will be assessed with a gas analyzer (Metalyzer 3B; CPX System, Leipzig, Germany), which will be calibrated before each test according to the manufacturer's recommendations. The gas analyzer will be calibrated with known concentrations of O2 and CO2 and the volume will be calibrated with a 3L syringe. Peak VO2 will be considered as the highest average values recorded in 10 seconds.
Anamnesis | It will only be performed before the intervention.
  The anamnesis will be conducted by applying a questionnaire prepared by the researcher as the initial stage of data collection, and contains questions involving personal information such as demographic aspects, self-reported skin color, education, marital status, number of people living in the household, family income, social vulnerability, polypharmacy, delirium, falls, incontinence, and presence of symptoms or clinical conditions detailed in the inclusion and exclusion criteria. In addition, information will be asked about history of physical exercise, type of work, injuries, surgery, family history of pathologies, time since HIV diagnosis (months), time of ARV use (months), therapies already administered, use of other medications, smoking, drugs, alcohol, co-infection with the Hepatitis C virus, whether the patient has suffered a stroke, chronic obstructive pulmonary disease, cardiovascular disease, and whether the patient has been diagnosed with COVID-19 (presence of sequelae).
Metabolic Parameters | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  To analyze the metabolic parameters of cardiovascular risks, serum levels of blood glucose (mg/dL), HDL-c (mg/dL), LDL-c (mg/dL), total cholesterol (mg/dL), and triglycerides (mg/dL) will be measured and evaluated. The analyses and collections will be performed at the Clinical Research Unit (UPC) of HC-FMRP/USP. The analyses will be performed using the enzymatic method using the Wiener Lab® Kit.
Height | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  It will be measured with the aid of an aluminum stadiometer, attached to the Filizola® brand electronic anthropometric scale, (Personal model for up to 180 kg, Campo Grande, MS), with a precision scale of 0.1 centimeters. The same scale used to measure body weight. The participant will remain in a static position, arms along the body, with bare feet. Keeping the head in the Frankfurt plane, and at the moment when the stadiometer accessory touches the upper part of the head of the person being assessed, forming a 90° angle, the measurement will be recorded.
Skinfold thicknesses | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The following regions will be measured accurately in mm: triceps, subscapular, suprailiac, horizontal abdominal, mid-thigh, and medial calf. The same skinfold caliper, made by Sanny®, Harpenden Scientific, with precision in mm and constant pressure of 10g/mm³, will be used for all measurements. The participant will remain standing, in a relaxed position, and the measurements will be taken in triplicate, with the median being recorded. If there is a variation greater than 5% between the measurements, a new series of measurements will be taken.
Body perimeters | From the beginning of recruitment to the end of the interventions will be approximately 15 weeks.
  The following regions will be measured with an accuracy of 0.1 centimeter: shoulder (largest diameter), chest (fourth costosternal joint), waist (smallest diameter), abdomen (umbilical scar), hip (largest diameter), extended right arm, flexed right arm, right forearm, right wrist, extended left arm, flexed left arm, left forearm, left wrist, right thigh (proximal), right calf (largest diameter), right ankle (smallest calf perimeter, closest to the malleoli), left thigh (proximal), left calf (largest diameter), and left ankle (smallest calf perimeter, closest to the malleoli). A 2-meter metal tape from the Sanny® brand will be used, with a latex device on the end. Measurements will be taken in triplicate, and the median will be recorded. If there is a variation greater than 5% between measurements, a new series of measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Andre P dos Santos, Professor Doutor, Study Director — University of Sao Paulo; Euripedes B G Gomide, Professor Doutor, Study Chair — Claretiano - Centro Universitário, Batatais, Brasil; Gianna F Marchiori, Doutora, Study Chair — Grupo de Pesquisa em Saúde Coletiva da Universidade Federal do Triângulo Mineiro, Uberaba, Brasil; Jéssica F C Cordeiro, Doutora, Study Chair — Faculdade de Desporto da Universidade do Porto, Porto, Portugal; Igor M Correia, Doutorando, Study Chair — University of Sao Paulo; Chimenny A L C de Moraes, Mestre, Study Chair — University of Sao Paulo; Alcivandro de S Oliveira, Mestrando, Study Chair — University of Sao Paulo; Camile V R de Oliveira, Graduada, Study Chair — University of Sao Paulo; Joana Brilhadori, Mestranda, Study Chair — University of Sao Paulo; Leandro C Nunes, Graduado, Study Chair — University of Sao Paulo; Lisa F Mazzonetto, Mestre, Study Chair — University of Sao Paulo; Jeferson R C dos Anjos, Mestre, Study Chair — University of Sao Paulo; Lara S Silva, Graduanda, Study Chair — Claretiano - Centro Universitário, Batatais, Brasil; Giovana Finco, Graduada, Study Chair — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: Yes
The raw data supporting the findings of this study will be available from the corresponding author upon reasonable notice.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code